CLINICAL TRIAL: NCT03677232
Title: The Living Experience of Hong Kong Chinese Adolescents With CHD.
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Other Study IDs: UW 17-290
Record Dates: First submitted 2018-09-05; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Congenital Heart Disease; Psychological Well-being; Quality of Life; Adolescent; Chinese
Keywords: Congenital Heart Disease, Hong Kong, Adolescent
MeSH Terms: conditions — Heart Defects, Congenital; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hong Kong Chinese adolescents with CHD: Hong Kong Chinese adolescents with CHD aged 12-18 who are able to read and write chinese

SUMMARY:
This study aims to explore the impacts of CHD and its limitations on adolescents and the living experience of adolescents living with CHD.

Hong Kong Chinese adolescents with CHD are having reduced psychological well-being and quality of life than their healthy counterparts. Qualitative study is therefore needed to explore how CHD may impact on the adolescents' psychological well-being and quality of life.

DETAILED DESCRIPTION:
A qualitative study was adopted. Purposive sampling of 30 adolescents with CHD were done. Thematic analysis was used for data analysis. The participants unfold negative impacts of CHD and its treatments, and the challenges they were facing with their relationship with others.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese adolescents
* aged 12 to 18
* able to read and write Chinese
* attending outpatient clinic of Department of Pediatric Cardiology

Exclusion Criteria:

* adolescents with non-structural heart disease
* with developmental delay or comorbid medical conditions

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hong Kong Chinese adolescents with CHD, aged 12 to 18, who are able to read and write Chinese, and are attending the outpatient clinic of Department of Pediatric Cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
living experience of adolescents with CHD | 1 day
  Participants were asked to describe their living experiences with CHD and how has CHD affected their quality of life and psychological well-being during the semi-structure interview.

CONTACTS AND LOCATIONS:
Overall Officials: William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No